CLINICAL TRIAL: NCT00405925
Title: Free Study: a Randomised, Open Label, Multicentre Strategic Study to Evaluate the Efficacy and Toxicity of an Early Switch From a PI-containing Regimen to Trizivir ® on Guidance of Viral Load in HIV-1 Infected , Antiretroviral naïve Adults
Brief Title: FREE Study: Efficacy and Toxicity of Trizivir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTC-184-010403
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: HIV Infections
Keywords: AIDS; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — abacavir, lamivudine, and zidovudine drug combination; Zidovudine; abacavir, lamivudine drug combination

ARMS (2):
- combivir/kaletra (Active Comparator): All patients started with combivir/Kaletra and were randomized if they reached undetectable viral load (2 times) within 24 weeks into continuation of the same regimen or Trizivir (2 arms)
  Interventions: Drug: zidovudine,lamivudine,abacavir
- Trizivir (Experimental): patients who reach undetectable HIV-RNA within 24 weeks are randomized to switch to trizivir or continuation of combivir/kaletra
  Interventions: Drug: Trizivir

INTERVENTIONS:
Drug: Trizivir
  Arms: Trizivir
Drug: zidovudine,lamivudine,abacavir — zidovudine 300 mg bid, lamivudine 150mg bid, abacavir 300mg bid
  Arms: combivir/kaletra

SUMMARY:
Antiretroviral naïve patients with <350 xE6/l CD4 cells and a HIV-viral load of > 30.000 cop/ml are started on combivir ® and Kaletra ®. When patients have reached an undetectable viral load of< 50 cop/ml on two consecutive occasions at least at week 12, but no later than week 24, they are randomised in either continuation with Combivir/Kaletra or switch to Trizivir ® twice daily one pill during 96 weeks. All patients randomised in the combivir/Kaletra arm are eligible to switch to Trizivir at any post randomisation visit when they reach predefined switch criteria for elevated levels of fasting glucose or lipids.

DETAILED DESCRIPTION:
The primary objective is to compare the antiviral efficacy of an early switch from a boosted PI/2NRTI regimen to Trizivir (after undetectability of HIV-RNA has been achieved on 2 consecutive occasions) with uninterrupted use of the PI/2NRTI regimen for 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age, confirmed HIV-1 infection, never received antiretrovirals before, plasma-HIV-RNA >30.000 cop/ml, CD4 < 350 E6/l.

Exclusion Criteria:

* pregnancy, women using proven barrier methods of contraception, defined uncontrolled active AIDS defining complication, being on treatment for diabetes, other serious illnesses, expected non-compliance, defined laboratory abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2003-03; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Plasma HIV-RNA < 400 cop/ml at week 96 for the Intent- To-Treat (ITT).

SECONDARY OUTCOMES:
HIV-RNA <50 cop at week 96
HIV-RNA <400 and <50 cop/ml at week 48
Time to virological failure
Immunological efficacy at week 48 and 96 measured by absolute change from baseline in CD4 cell counts
Duration of change in CD4 cell count from baseline to >200,
Proportion of subjects experiencing one or more predefined values of fasting glucose and triglycerides, LDL and LDL/HDL ratio
Development of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Richter, MD, Principal Investigator — Rijnstate Hospital, Arnhem, the Netherlands; P. Mulder, Study Director — Rijnstate Hospital, Arnhem, the Netherlands; N. Langebeek, Study Director — Rijnstate Hospital, Arnhem, the Netherlands; D. N. Burger, Study Director — Nijmegen, the Netherlands; P. P. Koopmans, Study Director — Nijmegen, the Netherlands; C. H. ten Napel, Study Director — Enschede, the Netherlands; P. H. Groeneveld, Study Director — Isala kliniek, Zwolle, the Netherlands; H. G. Sprenger, Study Director — Groningen, the Netherlands; R. W. ten Kate, Study Director — Haarlem, the Netherlands; M. E. van Kasteren, Study Director — Tilburg, the Netherlands; J. D. Le grand, Study Director — Charleroi, Belgium; R. Vriesendorp, Study Director — The Hague, the Netherlands; B. Bravenboer, Study Director — Eindhoven, the Netherlands; I. M. Hoepelman, Study Director — Utrecht, the Netherlands; P. van Bentum, Study Director — Rijnstate Hospital, Arnhem, the Netherlands; A. Smit-den Baars, Study Director — Rijnstate Hospital, Arnhem, the Netherlands
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands